CLINICAL TRIAL: NCT03620149
Title: Reduced Dose-density of Denosumab for Maintenance Therapy of Unresectable Giant Cell Tumor of Bone: a Multicenter Phase II Study "REDUCE"
Brief Title: Reduced Dose-density of Denosumab for Unresectable GCTB
Acronym: REDUCE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 1762-STBSG; 2018-002096-17 (EudraCT Number); 20177203 (Other: Amgen)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Bone Giant Cell Tumor
Keywords: denosumab; Giant cell tumor of bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Denosumab (Experimental): denosumab at reduced dose
  Interventions: Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA]

INTERVENTIONS:
Drug: Denosumab 120 MG/1.7 ML Subcutaneous Solution [XGEVA] — Denosumab 120 mg, SC, on day 1 of every 12-week cycle
  Other Names: Xgeva

SUMMARY:
This study is a multi-center, multi-national, open label, single arm phase 2 study of single-agent denosumab.

The objective of the trial is to evaluate the risk versus benefit of denosumab in maintenance setting in patients requiring long-term use (> 1 year) of denosumab. For that purpose, the treatment schedule with reduced dose density (120mg SC 12-weekly instead of 4-weekly) will be investigated, starting after 1-year (12-15 months) of denosumab full dose, as per current label. The impact on OsteoNecrosis of the Jaw (ONJ) without compromising disease control will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary or metastatic unresectable GCTB or resectable GCTB but not a candidate for surgery, excluding primary or metastatic GCTB in the jaw.
* Evidence of active disease at time of registration based on local investigator's assessment (according to RECIST v1.1)
* Age ≥ 18 years old and skeletally mature (ie, radiographic evidence of at least 1 mature long bone (e.g. humerus with closed growth epiphyseal plate)
* Patient must have received denosumab before entering this trial:
* The duration of treatment with full dose denosumab (120 mg SC ) as per current label must be at least 12 months and patient may have received up to 15 months of denosumab.
* And patient must have received at least 12 doses of denosumab 120 mg before entering into this trial.
* ECOG/WHO PS 0-2
* Albumin-adjusted serum calcium level ≥ 2.0 mmol/L (8.0 mg/dL)
* Representative formalin fixed, paraffin embedded tumor blocks or unstained tissue slides, either from the primary tumor or a metastatic lesion, must be available for histological central review.
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 7 days prior to the first reduced dose of study treatment.
* WOCBP should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 5 months after the last treatment cycle. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 5 months after the last study treatment.
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Currently receiving other GCTB specific treatment (eg, radiation, chemotherapy, or embolization)
* Concurrent bisphosphonate treatment and calcitonin
* Known or suspected current diagnosis of underlying malignancy including high-grade sarcoma, osteosarcoma, fibrosarcoma, malignant giant cell sarcoma
* Known diagnosis of second malignancy within the past 5 years (subjects with definitively treated basal cell carcinoma and cervical carcinoma in situ are permitted)
* Creatinine clearance < 30 mL/min
* Hemoglobin < 10.0 g/dL or 6.2 mmol/L
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw
* Active dental or jaw condition which requires oral surgery, including tooth extraction
* Non-healed dental/oral surgery
* Planned invasive dental procedure for the course of the study
* Known hypersensitivity to the active substance or to any of the excipients (glacial acetic acid, sodium hydroxide, sorbitol (E420), polysorbate 20)
* Treatment with other investigational device or drug 30 days prior to registration
* Known hypersensitivity to products to be administered during the study (calcium and/or vitamin D)
* Unstable systemic disease including active and uncontrolled infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months before registration
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 5.8 years after first patient in
  according to RECIST 1.1
Osteonecrosis of the jaw (ONJ) incidence | 5.8 years after first patient in

SECONDARY OUTCOMES:
Overall survival | 5.8 years after first patient in
Denosumab treatment duration | 5.8 years after first patient in
Occurrence of Adverse Events | 5.8 years after first patient in
  according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Palmerini, Study Chair — IRCCS Instituto Ortopedico Rizzoli; Hans Gelderblom, Study Chair — Leiden University Medical Center
Locations (8):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy
- Leiden University Medical Centre, Leiden, Netherlands
- Spain (4):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals (Institut Catala D'Oncologia), Barcelona
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Universitario San Carlos, Madrid
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
All publications must comply with the terms specified in the EORTC Policy 009 "Release of Results and Publication Policy".